CLINICAL TRIAL: NCT00486473
Title: Phase III Multicenter Double-Blind, Randomized, Crossover Study to Compare MultiHance With Magnevist in Contrast-enhanced Magnetic Resonance Imaging (MRI) of the Breast
Brief Title: Multihance Versus Magnevist in Breast MRI
Acronym: DETECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Gianpaolo Pirovano, M.D., Executive Director, Corporate Medical Development, Bracco Diagnostics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MH 131
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — gadobenic acid; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Multihance — 0.5 Molar at a single dose injection
Drug: Magnevist — 0.5M at a single dose injection

SUMMARY:
To show if one MRI contrast agent is better than another one in the diagnosis of malignant breast lesions compared to histopathology

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Female
* Age 18 years or older
* Suspicious or known breast lesion based on results from mammography or ultrasound
* Planned to undergo histological diagnosis of breast lesion by having a non surgical biopsy or breast surgery within 30 days after the MRI exam

Exclusion Criteria:

* Body weight > 100 kg
* Pregnant or lactating
* Server or end-stage organ failure
* Moderate to severe renal impairment
* Undergoing radiotherapy or completed radiotherapy in the last 18 months
* Chemotherapy within 6 months of the 1st MRI exam

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity in diagnosing breast lesions compared to histopathology results | up to 6 months

SECONDARY OUTCOMES:
Sensitivity, specificity, accuracy, PPV and NPV at region, breast and patient levels | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Dianostics, Inc.
Locations (1):
- Rome, Italy

REFERENCES:
- [Derived] Martincich L, Faivre-Pierret M, Zechmann CM, Corcione S, van den Bosch HC, Peng WJ, Petrillo A, Siegmann KC, Heverhagen JT, Panizza P, Gehl HB, Diekmann F, Pediconi F, Ma L, Gilbert FJ, Sardanelli F, Belli P, Salvatore M, Kreitner KF, Weiss CM, Zuiani C. Multicenter, double-blind, randomized, intraindividual crossover comparison of gadobenate dimeglumine and gadopentetate dimeglumine for Breast MR imaging (DETECT Trial). Radiology. 2011 Feb;258(2):396-408. doi: 10.1148/radiol.10100968. Epub 2010 Dec 16. PMID 21163915